CLINICAL TRIAL: NCT00629824
Title: Efficacy and Safety of Pegylated Interferon Plus Ribavirin Combination Therapy in Treating Older Patients With Chronic Hepatitis C
Brief Title: Pegylated Interferon Plus Ribavirin in Treating Older Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Ming-Lung Yu, Kaohsiung Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB- 960047
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; sustained virological response; rapid virological response; peginterferon; ribavirin; old age
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): 110 naïve CHC patients who are 65 to 80 years of age
  Interventions: Drug: pegylated interferon alpha and plus ribavirin
- B (Active Comparator): 140 naïve CHC patients who are 50 to 64 years of age
  Interventions: Drug: pegylated interferon alpha and plus ribavirin
- C (Active Comparator): 40 HCV-1 infected patients with an RVR who are 65-80 years of age will receive 24 weeks of treatment
  Interventions: Drug: pegylated interferon alpha and plus ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha and plus ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day, 24weeks of treatment for genotype non-1 infected patients and 48 weeks of treatment for genotype 1 infected patients, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: A
Drug: pegylated interferon alpha and plus ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day, 24weeks of treatment for genotype non-1 infected patients and 48 weeks of treatment for genotype 1 infected patients, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: B
Drug: pegylated interferon alpha and plus ribavirin — pegylated interferon alpha 180 ug/week and ribavirin 1000-1200 mg/day for 24 weeks
  Other Names: PEGASYS®
  Arms: C

SUMMARY:
Combination therapy with pegylated interferon-alpha plus ribavirin has greatly improved the treatment efficacy and is the mainstream of treatment for chronic hepatitis C infection. The efficacy and safety of pegylated interferon-alpha plus ribavirin combination therapy and its impact on the outcome in older patients with chronic hepatitis C deserve to be elucidated.

The purposes of this study are:

1. To evaluate the efficacy of pegylated interferon-alpha 2a plus ribavirin combination therapy in older patients with chronic hepatitis C
2. To investigate the safety of pegylated interferon-alpha 2a plus ribavirin combination therapy in older patients with chronic hepatitis C

DETAILED DESCRIPTION:
A prospective, hospital-based, case-control study enrolling 70 chronic hepatitis C patients who are 65 to 80 years of age and other sex- and HCV genotype-matched 140 chronic hepatitis C patients who are 50 to 64 years of age will be conducted for comparison. The 210 patients chronic hepatitis C patients will receive pegylated interferon-alpha plus ribavirin combination therapy. Genotype 1 infected patients will received 48 weeks of treatment and genotype non-1 patients will received 24 weeks of treatment. Another 40 HCV-1 infected patients who are 65-80 years of age and have a rapid virological response ( defined as seronegative of HCV RNA at week 4 of treatment) will receive 24 weeks of treatment and are enrolled for comparison since Jan 2008. The primary outcome measurement is sustained virological response and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >50 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Present therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Clinical evidence or history of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption>40 g/day) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb <11 g/dL in women or <12 g/dL in men at screening
* Any patient with major thalassemia
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* Local or Systemic malignancy unstable status

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period. | 1.5 year

SECONDARY OUTCOMES:
RVR, rapid virological response, defined as HCV RNA < 50 IU/mL at treatment week 4 | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD, PhD, Principal Investigator — Kaohsiung Medical University; Jee-Fu Huang, MD, Principal Investigator — Kaohsiung Municipal Hsiao-Kang Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Antonucci G, Longo MA, Angeletti C, Vairo F, Oliva A, Comandini UV, Tocci G, Boumis E, Noto P, Solmone MC, Capobianchi MR, Girardi E. The effect of age on response to therapy with peginterferon alpha plus ribavirin in a cohort of patients with chronic HCV hepatitis including subjects older than 65 yr. Am J Gastroenterol. 2007 Jul;102(7):1383-91. doi: 10.1111/j.1572-0241.2007.01201.x. Epub 2007 Mar 31. PMID 17403072
- [Background] Hiramatsu N, Oze T, Tsuda N, Kurashige N, Koga K, Toyama T, Yasumaru M, Kanto T, Takehara T, Kasahara A, Kato M, Yoshihara H, Katayama K, Hijioka T, Hagiwara H, Kubota S, Oshita M, Haruna Y, Mita E, Suzuki K, Ishibashi K, Hayashi N. Should aged patients with chronic hepatitis C be treated with interferon and ribavirin combination therapy? Hepatol Res. 2006 Jul;35(3):185-9. doi: 10.1016/j.hepres.2006.03.008. Epub 2006 May 4. PMID 16678478
- [Background] Thabut D, Le Calvez S, Thibault V, Massard J, Munteanu M, Di Martino V, Ratziu V, Poynard T. Hepatitis C in 6,865 patients 65 yr or older: a severe and neglected curable disease? Am J Gastroenterol. 2006 Jun;101(6):1260-7. doi: 10.1111/j.1572-0241.2006.00556.x. PMID 16771947
- [Background] Honda T, Katano Y, Urano F, Murayama M, Hayashi K, Ishigami M, Nakano I, Yoshioka K, Toyoda H, Kumada T, Goto H. Efficacy of ribavirin plus interferon-alpha in patients aged >or=60 years with chronic hepatitis C. J Gastroenterol Hepatol. 2007 Jul;22(7):989-95. doi: 10.1111/j.1440-1746.2006.04773.x. PMID 17608843
- [Background] Iwasaki Y, Ikeda H, Araki Y, Osawa T, Kita K, Ando M, Shimoe T, Takaguchi K, Hashimoto N, Kobatake T, Tomita M, Kawaguchi M, Kobashi H, Sakaguchi K, Shiratori Y. Limitation of combination therapy of interferon and ribavirin for older patients with chronic hepatitis C. Hepatology. 2006 Jan;43(1):54-63. doi: 10.1002/hep.20984. PMID 16374855
- [Derived] Huang CF, Yang JF, Dai CY, Huang JF, Hou NJ, Hsieh MY, Lin ZY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL, Yu ML. Efficacy and safety of pegylated interferon combined with ribavirin for the treatment of older patients with chronic hepatitis C. J Infect Dis. 2010 Mar;201(5):751-9. doi: 10.1086/650470. PMID 20102281